CLINICAL TRIAL: NCT07155135
Title: Magnetic Resonance Imaging Safety in Patients With Non-Conditional, Mixed-Manufacturer Cardiac Implantable Electronic Devices
Brief Title: Safety of Magnetic Resonance Imaging With Patients Who Have Mixed Lead Cardiac Implantable Electronic Devices
Acronym: MRIMLD
Status: Completed | Type: Observational
Sponsor: Socal Heart (Industry)
Responsible Party: Principal Investigator, Ryka Tashakkor, First Author, Socal Heart
Other Study IDs: 2025818
Record Dates: First submitted 2025-08-19; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Safety of MRI
Keywords: cardiac implantable electronic devices; CIED; MRI; Magnetic Resonance Imaging; safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with mixed-lead Cardiac Implantable Electronic Devices: Patients recieved clinical relevant MRI's. Patients are checked for complications post-MRI.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Magnetic resonance imaging (MRI) is a vital diagnostic tool in modern medicine due to its ability to produce detailed images of the body's internal structures without using ionizing radiation.

SUMMARY:
This study is looking at the safety and efficacy of using MRIs with patients who have cardiac implantable electronic devices.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) is a critical diagnostic tool known for its non-invasive nature and high-resolution imaging capabilities. However, its safety in patients with cardiac implantable electronic devices (CIEDs), particularly those with mixed-lead systems, remains a significant clinical concern. This report investigates the safety and efficacy of MRI in such patients, where generators and leads originate from different manufacturers and are not officially deemed MRI-conditional.

ELIGIBILITY:
Inclusion Criteria:

* have a mixed-lead CIED
* clinical relevant MRI

Exclusion Criteria:

* same manufactured CIED

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Average age of patients are 82 years old. All 100% of RA leads and devices were manufactured by Abbott; 31% of RV leads were manufactured by Boston Scientific, with the remaining 69% of RV leads by Medtronic.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Evaluation of Changes in Device Battery Voltage (Volts) | Immediately Prior to MRI and Immediately after MRI
  report Device Battery Voltage (in Volts) prior to the MRI and after the MRI and determine if there was a change in voltage greater than 10% from the initial measurement to the final measurement.
Evaluation of Changes in Lead Impedance (Ohms) | Immediately Prior to MRI and Immediately after MRI
  report lead impedance (in Ohms) prior to the MRI and after the MRI and determine if there is a change in impedence greater than 20% from the initial measurement to the final measurement.
Evaluation of Changes in Lead Threshold (Voltage) Before and After MRI | Immediately Prior to MRI and Immediately after MRI
  report lead threshold in (voltage) prior to MRI and after the MRI and determine if there is a change greater than10% from the initial measurement to the final measurement.

SECONDARY OUTCOMES:
Evaluation of Changes in Patient Clinical Outcomes (Rhythm, Symptoms, Cardiac Arrest, or Death) Before and After MRI | Immediately Prior to MRI and Immediately after MRI
  We will review medical records and determine if there were any observed change in patient rhythm, symptoms (such as chest pain, syncope), cardiac arrest or death after the MRI was completed.

CONTACTS AND LOCATIONS:
Overall Officials: Babak Tashakkor, MD, Study Director — Southern California Heart Specialists
Locations (1):
- Southern California Heart Specialists, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy.

REFERENCES:
- [Result] Russo RJ, Costa HS, Silva PD, Anderson JL, Arshad A, Biederman RW, Boyle NG, Frabizzio JV, Birgersdotter-Green U, Higgins SL, Lampert R, Machado CE, Martin ET, Rivard AL, Rubenstein JC, Schaerf RH, Schwartz JD, Shah DJ, Tomassoni GF, Tominaga GT, Tonkin AE, Uretsky S, Wolff SD. Assessing the Risks Associated with MRI in Patients with a Pacemaker or Defibrillator. N Engl J Med. 2017 Feb 23;376(8):755-764. doi: 10.1056/NEJMoa1603265. PMID 28225684
- [Result] Nazarian, S., Hansford, R., Rahsepar, A. A., et al. (2021). "MRI for patients with non-MRI-conditional cardiac devices." The New England Journal of Medicine, 384(7), 674-675.
- [Result] Russo, R. J., Costa, H. S., Silva, P. D., et al. (2017). "Assessing the risks associated with MRI in patients with cardiac devices." Journal of the American College of Cardiology, 69(8), 1123-1133.
- [Result] Lanz H, Strauss K, Hopler J, Kraft M, Hoffmann S, Binzenhofer L, Gade N, Roden D, Saleh I, Kaab S, Lackermair K, Sadoni S, Hagl C, Massberg S, Estner H, Fichtner S, Lusebrink E. Safety of Magnetic Resonance Imaging in Patients with Cardiac Implantable Electronic Devices. J Cardiovasc Dev Dis. 2024 Oct 8;11(10):313. doi: 10.3390/jcdd11100313. PMID 39452284
- [Result] Nazarian S, Hansford R, Rahsepar AA, Weltin V, McVeigh D, Gucuk Ipek E, Kwan A, Berger RD, Calkins H, Lardo AC, Kraut MA, Kamel IR, Zimmerman SL, Halperin HR. Safety of Magnetic Resonance Imaging in Patients with Cardiac Devices. N Engl J Med. 2017 Dec 28;377(26):2555-2564. doi: 10.1056/NEJMoa1604267. PMID 29281579
- [Result] Mason S, Osborn JS, Dhar R, Tonkin A, Ethington JD, Le V, Benuzillo J, Lappe DL, Knowlton KU, Bunch TJ, Anderson JL. Real world MRI experience with nonconditional and conditional cardiac rhythm devices after MagnaSafe. J Cardiovasc Electrophysiol. 2017 Dec;28(12):1468-1474. doi: 10.1111/jce.13351. Epub 2017 Nov 1. PMID 28960745
- [Result] Martin ET, Sandler DA. MRI in patients with cardiac devices. Curr Cardiol Rep. 2007 Mar;9(1):63-71. doi: 10.1007/s11886-007-0012-y. PMID 17362687
- [Result] Madigan JD, Choudhri AF, Chen J, Spotnitz HM, Oz MC, Edwards N. Surgical management of the patient with an implanted cardiac device: implications of electromagnetic interference. Ann Surg. 1999 Nov;230(5):639-47. doi: 10.1097/00000658-199911000-00005. PMID 10561087
- [Result] Driller J, Barold SS, Parsonnet V. Normal and abnormal function of the pacemaker magnetic reed switch. J Electrocardiol. 1976;9(3):283-92. doi: 10.1016/s0022-0736(76)80058-1. PMID 781163
- [Result] Irnich W, Irnich B, Bartsch C, Stertmann WA, Gufler H, Weiler G. Do we need pacemakers resistant to magnetic resonance imaging? Europace. 2005 Jul;7(4):353-65. doi: 10.1016/j.eupc.2005.02.120. PMID 15944094
- [Result] Luechinger R, Zeijlemaker VA, Pedersen EM, Mortensen P, Falk E, Duru F, Candinas R, Boesiger P. In vivo heating of pacemaker leads during magnetic resonance imaging. Eur Heart J. 2005 Feb;26(4):376-83; discussion 325-7. doi: 10.1093/eurheartj/ehi009. Epub 2004 Nov 29. PMID 15618060
- [Result] Kodali S, Baher A, Shah D. Safety of MRIs in patients with pacemakers and defibrillators. Methodist Debakey Cardiovasc J. 2013 Jul-Sep;9(3):137-41. doi: 10.14797/mdcj-9-3-137. PMID 24066196
- [Result] Luechinger R, Duru F, Scheidegger MB, Boesiger P, Candinas R. Force and torque effects of a 1.5-Tesla MRI scanner on cardiac pacemakers and ICDs. Pacing Clin Electrophysiol. 2001 Feb;24(2):199-205. doi: 10.1046/j.1460-9592.2001.00199.x. PMID 11270700
- [Result] Ferreira AM, Costa F, Tralhao A, Marques H, Cardim N, Adragao P. MRI-conditional pacemakers: current perspectives. Med Devices (Auckl). 2014 May 7;7:115-24. doi: 10.2147/MDER.S44063. eCollection 2014. PMID 24851058
- See also: MagnaSafe Registry. Summary of the MagnaSafe Protocol. — http://www.cms.gov/medicare-coverage-database/view/ncacal-decision-memo.aspx?NCAId=289&proposed=N&utm
- See also: University of Wisconsin-Madison. MRI Safety Subcommittee on Pacemakers: 2018 Revision. Madison (WI): University of Wisconsin-Madison, Department of Radiology — https://www.radiology.wisc.edu/wp-content/uploads/2018/11/MRI_Safety_Subcomittee_on_Pacemakers_Memo_2018rev.pdf
- See also: Initial data presented on world's first MRI-safe pacemaker. DAIC DiCardiology. 2008 Sep 1 [cited 2025 Jun 21] — https://www.dicardiology.com/content/initial-data-presented-worlds-first-mri-safe-pacemaker
- See also: MRI Safety in Patients with Cardiac Implantable Electronic Devices: A Review. Radiology. 2018 — https://s.mriquestions.com/uploads/3/4/5/7/34572113/muthalalyradiol.2018180285.pdf